CLINICAL TRIAL: NCT00077883
Title: Phase 1-2a Dose-Ranging Study of TLK286 in Combination With Cisplatin as First-Line Therapy in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: TLK286 (Telcyta) in Combination With Cisplatin for Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, MD Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2021
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2005-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TER 286; Cisplatin

INTERVENTIONS:
Drug: TLK286, cisplatin — TLK286 administered once every 3 weeks (± 2 days) at two dose-ranging levels (750 mg/m²) and 1,000 mg/²) in combination with two dose levels of cisplatin (75 mg/m² and 100 mg/m²) of cisplatin once every 3 weeks (± 2 days).

SUMMARY:
The purpose of this trial is to study the efficacy and safety of the combination of TLK286 with cisplatin as first-line therapy for patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed non-small cell lung cancer
* Stage IV or IIIB
* Measurable disease by RECIST
* ECOG performance status of 0-1
* Adequate liver and renal function
* Adequate bone marrow reserve

Exclusion Criteria:

* History of bone marrow transplantation or stem cell support
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Primary Objectives of the Study | Every 3 weeks
  1. To determine the safety of TLK286 in combination with cisplatin in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC)
  2. To determine the MTD of TLK286 in combination with cisplatin in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Univ. of MD, Greenbaum Cancer Center, Baltimore, Maryland
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Univ. of TX, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Related Info — http://www.telik.com